CLINICAL TRIAL: NCT00200278
Title: Exercise Instruction Via Phone or Print
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: Brown University (Other); Stanford University (Other); University of Pittsburgh (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: R01HL064342 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-09

CONDITIONS: Cardiovascular Disease
Keywords: Exercise; Intervention studies; Decision-making; computer assisted Expert systems; telephone
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity

INTERVENTIONS:
Behavioral: PROJECT STRIDE

SUMMARY:
The objective of this study is to determine the differential effect of intervention delivery channel (phone versus print versus wait list control) on physical activity adoption and maintenance in previously sedentary adults. Both delivery channels have been found to be effective, but telephone-based interventions require more commitment on the part of the subjects and are more labor intensive than print-based interventions. Thus, we will conduct a randomized controlled clinical trial comparing three groups: 1) telephone-based motivationally-tailored individualized feedback; 2) print-based, motivationally-tailored individualized feedback; 3) minimal contact waiting list control condition (receive intervention after 12 months as controls). Two hundred and twenty-eight healthy, sedentary women and men ages 18-65 will be randomly assigned to one of the two interventions or the waiting-list control condition. Our primary hypothesis is that individuals randomized to either phone or print conditions will exhibit significantly higher levels of physical activity participation at 6 and 12 months than individuals in the waiting list control condition. And, in addition, that subjects randomized to the telephone condition will exhibit significantly higher levels of physical activity participation at 6 and 12 months than those in the print condition.

DETAILED DESCRIPTION:
As many as 60% of Americans do not engage in regular physical activity and 25% are completely inactive. The risk of cardiovascular disease is almost doubled among people who are physically inactive, comparable to the risks associated with increased systolic blood pressure, cigarette smoking, and elevated serum cholesterol. To make an impact on physical activity prevalence at the population level requires a research focus at the interface between clinical efficacy trials and large-scale dissemination studies. Studies at this interface must use proven interventions that are simultaneously effective and cost-efficient. Such interventions are the focus of this proposal.

The objective of this study is to determine the differential effect of intervention delivery channel (phone versus print versus wait list control) on physical activity adoption and maintenance in previously sedentary adults. Both delivery channels have been found to be effective, but telephone-based interventions require more commitment on the part of the subjects and are more labor intensive than print-based interventions. Thus, we will conduct a randomized controlled clinical trial comparing three groups: 1) telephone-based motivationally-tailored individualized feedback; 2) print-based, motivationally-tailored individualized feedback; 3) minimal contact waiting list control condition (receive intervention after 12 months as controls). Two hundred and twenty-eight healthy, sedentary women and men ages 18-65 will be randomly assigned to one of the two interventions or the waiting-list control condition. The two intervention arms will be matched with respect to frequency and content of contact. Data will be collected at baseline, 6, and 12 months using well-established physical activity and physical performance measures, as well as a comprehensive set of psychosocial questionnaires. Our primary hypothesis is that individuals randomized to either phone or print conditions will exhibit significantly higher levels of physical activity participation at 6 and 12 months than individuals in the waiting list control condition. And, in addition, that subjects randomized to the telephone condition will exhibit significantly higher levels of physical activity participation at 6 and 12 months than those in the print condition. Additional questions of interest include evaluation of the cost-effectiveness of the two intervention delivery approaches, each in relation to each other and to the wait list control group and examination of potential moderators and mediators of the intervention-physical activity relationship. This study will contribute important information regarding the relative efficacy and cost-effectiveness of two interventions, each of which can be utilized for widespread public health dissemination.

ELIGIBILITY:
Inclusion Criteria:

Individuals between the ages of 18 to 65 years were recruited for this study. Criteria for study participation were that individuals were healthy and under-active (i.e., participating in moderate or vigorous physical activity for 90 minutes or less per week).

Exclusion Criteria:

Individuals were excluded from the study if their body mass index (BMI) was greater than 35 or if they had hypertension, heart disease of any kind or an abnormal electrocardiogram, stroke, chronic infectious disease, any musculoskeletal problem which would limit treadmill testing or impair their ability to exercise, asthma, emphysema, chronic bronchitis, or any other serious medical condition that might make exercise unsafe or unwise. Other exclusion criteria were a schedule that would make adherence unlikely (such as very frequent travel), plans to move from the area within the next year, pregnancy or plans to attempt pregnancy, self-report of more than three alcoholic drinks per day on 5 or more days per week, hospitalization for a psychiatric disorder within the last 6 months, currently suicidal, bipolar, or psychotic, or currently using prescription medication that might impair exercise performance or tolerance, specifically beta blockers. Participants agreed to be randomly assigned to any of the conditions and read and signed an institutionally approved consent form after all their questions were answered.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 228
Dates: Start 2000-08; Study Completion 2005-03

PRIMARY OUTCOMES:
7 day Physical Activity Recall

SECONDARY OUTCOMES:
Exercise Stages of Change
Estimated VO2 max
Treadmill time

CONTACTS AND LOCATIONS:
Overall Officials: Bess H Marcus, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- Centers for Behavioral and Preventive Medicine/Miriam Hospital, Providence, Rhode Island, United States